CLINICAL TRIAL: NCT01741298
Title: Biobehavioral Bases & Management of Metabolic Syndrome
Brief Title: Biobehavioral Bases & Management of Metabolic Syndrome (CHARMS)
Acronym: CHARMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Neil Schneiderman, Professor, University of Miami
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P01 HL 36588- Proj 2; P01HL036588 (NIH)
Record Dates: First submitted 2012-11-27; First posted 2012-12-04 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle counseling (Experimental): CHARMS Intervention Participants (Pts) randomized to the lifestyle intervention received a yr long, 17 session intervention. Pts were asked to wear a pedometer and record their food intake for at least the week prior to each session. The first 4 sessions were delivered weekly, followed by 4 sessions delivered biweekly and finally 9 sessions delivered monthly. Each session was approximately 1-2 hrs. At the beginning of each session anthropometric, physical activity and dietary data were collected. Participants were lead in a 5 min deep breathing exercise before the didactic portion of the session began. Sessions targeted a broad range of material related to diet, physical activity, and psychosocial well-being. Participants were given homework assignments to incorporate covered material into their daily lives. Participants randomized to the intervention arm received follow-up assessments at 6 and 12 months post randomization.
  Interventions: Behavioral: CHARMS

INTERVENTIONS:
Behavioral: CHARMS — Participants (Pts) randomized to the lifestyle intervention received a yr long, 17 session intervention. Pts were asked to wear a pedometer and record their food intake for at least the week prior to each session. The first 4 sessions were delivered weekly, followed by 4 sessions delivered biweekly and finally 9 sessions delivered monthly. Each session was approximately 1-2 hrs. At the beginning of each session anthropometric, physical activity and dietary data were collected. Participants were lead in a 5 min deep breathing exercise before the didactic portion of the session began. Sessions targeted a broad range of material related to diet, physical activity, and psychosocial well-being. Participants were given homework assignments to incorporate covered material into their daily lives. Participants randomized to the intervention arm received follow-up assessments at 6 and 12 months post randomization.

SUMMARY:
The metabolic syndrome is increasingly being recognized as a major threat to good health - especially cardiovascular health - and its frequency appears to be increasing in relation to the current epidemic of obesity. The objective of this study is to determine whether a program of enhanced lifestyle intervention can, compared to standard care, reduce the frequency and severity of the metabolic syndrome as assessed by clinical, metabolic, inflammatory and vascular outcome measures. EC will consist of a 17-session structured, lifestyle intervention plan, directed at achieving weight reduction and increasing physical activity change through education, behavior modification and stress management, and conducted in groups. It will comprise a 3-month Core Curriculum of 8 sessions, followed by a Maintenance phase with 9 monthly sessions delivered by lifestyle counselors, experienced in breaking through barriers in working with socioeconomically disadvantaged members of minority groups. All participants will have baseline, 6-monthly and 1-year assessments. This project, Project 2, entitled Community Health Approaches to Reducing Risk in the Metabolic Syndrome (CHARMS), seeks to study psychosocial and behavioral (lifestyle) variables that may contribute to the progression or amelioration of atherosclerotic processes underlying the pathogenesis of coronary heart disease (CHD).

DETAILED DESCRIPTION:
The metabolic syndrome is increasingly being recognized as a major threat to good health - especially cardiovascular health - and its frequency appears to be increasing in relation to the current epidemic of obesity. The objective of this study is to determine whether a program of enhanced lifestyle intervention can, compared to standard care, reduce the frequency and severity of the metabolic syndrome as assessed by clinical, metabolic, inflammatory and vascular outcome measures. The project will compare the effects of Enhanced Care (EC) in 112 patients (80 completers) to Standard Care (SC) in 112 patients (80 completers) over a 12-month period. Following 3 run-in sessions given to both SC and EC participants, eligible subjects randomized to SC will receive lifestyle modification advice as recommended management of the metabolic syndrome and this will be administered at the baseline and the 6 month assessment visits. EC will consist of a 17-session structured, lifestyle intervention plan, directed at achieving weight reduction and increasing physical activity change through education, behavior modification and stress management, and conducted in groups. It will comprise a 3-month Core Curriculum of 8 sessions, followed by a Maintenance phase with 9 monthly sessions delivered by lifestyle counselors, experienced in breaking through barriers in working with socioeconomically disadvantaged members of minority groups. All participants will have baseline, 6-monthly and 1-year assessments. This project, Project 2, entitled Community Health Approaches to Reducing Risk in the Metabolic Syndrome (CHARMS), seeks to study psychosocial and behavioral (lifestyle) variables that may contribute to the progression or amelioration of atherosclerotic processes underlying the pathogenesis of coronary heart disease (CHD). Outcome variables will include measures of glycemic control/insulin resistance and/or dyslipidemia, oxidative stress, inflammation and overt manifestations of disease.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age 30-70 years
* Language: English or Spanish
* At least 3 features of the NCEP ATP-III metabolic syndrome

Exclusion Criteria:

* Diabetes
* Established CVD
* Uncontrolled hypertension (systolic BP >160 and diastolic BP >100 mm Hg)
* Established liver disease
* Renal insufficiency
* Psychiatric illness
* Chronic substance abuse within the past 5 years
* Chronic obstructive pulmonary disease or severe asthma.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2008-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Weight loss | 1 year
  Weight will be checked during each intervention session with the goal of losing 7% of total body weight from the enrollment date.

SECONDARY OUTCOMES:
Measures of glycemic control/insulin resistance. | 1 year
  Secondary outcomes measures will include glycemic control aka insulin resistance.

REFERENCES:
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717